CLINICAL TRIAL: NCT03762239
Title: Citizen Science for Analysing the Effect of Air Pollution on the Cognitive Function of Adolescents
Brief Title: Effect of Air Pollution on the Cognitive Function of Adolescents
Acronym: ATENC!Ó
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barcelona Institute for Global Health (Other)
Collaborators: Recercaixa (Unknown); Centre de Recerca per a l'Educació Científica i Matemàtica (CRECIM) (Unknown); Institute of Environmental Assessment and Water Research (IDAEA-CSIC) (Unknown); Economics and Bussiness Department, Universtitat Pompeu Fabra (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PI2030
Record Dates: First submitted 2018-11-23; First posted 2018-12-03 (Actual); Results first posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Attention Impaired; Risk-Taking; Risk Behavior; Social Preferences; Decision Making; Attention
Keywords: Attention; Air pollution; Black carbon; Particulate matter; Risk behavior; Social preferences; Decision making; Air purifier; Air cleaner
MeSH Terms: conditions — Risk-Taking | interventions — Air Filters

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Purified air (Active Comparator): Purifying the air with a Pure Airbox device (Zonair 3D). Use of air purifier (Pure Airbox, Zonair 3D) in the classroom 30 minutes before the participants enter the room and during the 2 hours of the experiment.
  Interventions: Other: Purifying the air with a Pure Airbox device (Zonair 3D)
- Normal air (Sham Comparator): Using a sham air purifier (same device without filters). Use of the same air purifier but without filters, so that it only recirculates the air without purifying it. Used for the same time period than the other arm.
  Interventions: Other: Using a sham air purifier (same device without filters)

INTERVENTIONS:
Other: Purifying the air with a Pure Airbox device (Zonair 3D) — Purifying the air of the classroom where the experiment is conducted using a Pure Airbox device (Zonair 3D)
  Other Names: Air filtering; Air cleaning
  Arms: Purified air
Other: Using a sham air purifier (same device without filters) — Use the air purifier (Pure Airbox, Zonair 3D) without filters in the classroom where the experiment is conducted
  Other Names: Sham air cleaner
  Arms: Normal air

SUMMARY:
Previous observational studies have reported an association between higher air pollution exposure and lower attention in children. With this project, the investigators aim to confirm this association in adolescents using an experimental design. In addition, the study will assess the relationship between air pollution exposure and individual preferences with respect to risk, time and social considerations. High school students in 3rd grade (ESO, 14-15 years of age) in different high schools in the Barcelona province (Spain) will be invited to participate. For each class in each high school, participating students will be randomly split into two equal-sized groups. Each group will be assigned to a different classroom where they will complete several activities during two hours, including an attention test (Flanker task) and a reduced version of the Global Preferences Survey. One of the classrooms will have an air purifier that will clean the air. The other classroom will have the same device but without the filters, so it will only re-circulate the air without cleaning it. Students will be masked to intervention allocation. The investigators hypothesize that students assigned to the clean air classroom will have better scores in the attention test, and that decision-making will also present differences in the two classrooms.

ELIGIBILITY:
Inclusion Criteria:

* Students in the 3rd ESO course in participating high schools with signed informed consent

Exclusion Criteria:

* None

Ages: 13 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2123 (Actual)
Dates: Start 2018-11-23 (Actual); Primary Completion 2019-06-11 (Actual); Study Completion 2019-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Basagaña, PhD, Principal Investigator — Barcelona Institute for Global Health
Locations (1):
- ISGlobal, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD except identifying information for participants or high schools will be shared
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will become available when publishing the results in a scientific journal, with no time restrictions
Access Criteria: Access to anyone via a public repository

RESULTS

PARTICIPANT FLOW:
Recruitment Details: To recruit participants (students), the objectives and design of the study were presented during teacher training sessions opened to all science teachers from all high schools of Barcelona metropolitan area. Teachers interested in participating signed up in an online form. Teachers from 33 high schools reached out to the research team to participate.
Pre-assignment Details: Based on 33 participating high schools, 2670 students were estimated eligible. As the total number of eligible students was not retrieved at the onset of the study, this estimation was based on the maximum number of students per class (n = 30), and thus it was likely to be overestimated. Of these, 547 individuals were excluded prior to randomization (parents or legal guardians who did not sign the consent form or students who declined to participate).
Period: Overall Study
Arm/Group | Purified Air | Normal Air
Started | 1068 | 1055
Completed | 1067 | 1054
Not Completed | 1 | 1
Not completed — Appointment to the doctor | 1 | 1

BASELINE CHARACTERISTICS:
Population: Students not having completed both ANT tests or showing low accuracy were excluded from the main analysis. An ANT test was considered a low accuracy test when the number of correct responses was less than 70%. Thus, a total of 68 participants from purified air group and 60 from normal air group were excluded from analysis (analytical sample, N = 1993)
Groups:
- Total: Total of all reporting groups
Arm/Group | Purified Air | Normal Air | Total
Number analyzed (Participants) | 999 | 994 | 1993
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 14.7 [14.6 to 14.8] | 14.7 [14.6 to 14.9] | 14.7 [14.6 to 14.9]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex: Female | 514 | 483 | 997
  Sex: Male | 481 | 507 | 988
  Sex: Other | 4 | 4 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
PMA-R, Primary Mental Aptitudes - Reasoning [Median (Inter-Quartile Range); unit: score] — Scale from 0 to 20 and lower values represent a worse outcome
  score | 17 [12 to 20] | 16 [11 to 20] | 16 [12 to 20]
HRT-SE, hit reaction time standard error [Median (Inter-Quartile Range); unit: ms] — HRT-SE represents the response speed consistency. The measure is calculated as hit reaction time (in ms) standard error for correct responses (HRT-SE). A lower HRT-SE indicates consistent reaction times and thus, a better attention performance.
  ms | 164.1 [114.5 to 237.3] | 158.6 [110.7 to 238.5] | 161.7 [112.6 to 237.9]
Impulsivity [Median (Inter-Quartile Range); unit: total score] — Impulsivity represents the number of incorrect responses (responses made in the opposite direction to the direction of the target arrow). Total range score is: 0-38. Higher values represent a worse outcome.
  total score | 2 [1 to 3] | 2 [1 to 3] | 2 [1 to 3]
Selective attention [Median (Inter-Quartile Range); unit: total score] — The number of omission errors (failure to respond to the stimulus). Total range score : 0-21. Higher values represent a worse outcome
  total score | 0 [0 to 1] | 0 [0 to 0] | 0 [0 to 0]
Alerting [Median (Inter-Quartile Range); unit: ms] — Alerting is computed by subtracting the median reaction time for double cue from median reaction time for the no cue condition (calculations performed after removing the incongruent trials). Higher values represent a worse outcome
  ms | 34.5 [5 to 66] | 35.5 [10 to 64.5] | 34.5 [7.5 to 65.5]
Orienting [Median (Inter-Quartile Range); unit: ms] — Orienting is computed by subtracting the median reaction time for spatial cue from the reaction time for central cue (calculations performed after removing the incongruent trials). Higher values represent a worse outcome
  ms | 14 [-12 to 40] | 14.8 [-9 to 40.5] | 14 [-10.5 to 40]
Conflict [Median (Inter-Quartile Range); unit: ms] — Conflict generally refers to the ability to monitor and resolve conflict among responses and in this study it is calculated as the median reaction time for each flanker condition (across cue conditions) and subtracting the congruent from the incongruent reaction times. Higher values represent a worse outcome
  ms | 78 [58.5 to 100] | 76.5 [56 to 97.5] | 77 [57.5 to 98.5]

OUTCOME MEASURES:

1. Primary Outcome: Response Speed Consistency Throughout the Attention Network Task-Flanker Task (Post ANT)
Description: This is a measure related to attentiveness that is calculated as hit reaction time standard error for correct responses (HRT-SE).
  A higher HRT-SE indicates highly variable reactions during the ANT test that is related to inattentiveness.
  A lower HRT-SE indicates indicates consistent reaction times and thus, a better attention performance.
Time Frame: Obtained from a test administered approximately 90 minutes after entering the classroom
Measure: Median (Inter-Quartile Range); unit: ms
Arm/Group | Purified Air | Normal Air
Number analyzed (Participants) | 999 | 994
ms | 161.3 [112.7 to 232.4] | 160.2 [112.4 to 234.7]
Statistical Analysis 1: Comparison: Purified Air vs Normal Air; The hypothesis was that air filtration could result in better performance, relative to the classroom without air filter (normal air), in attention measures among adolescents in high schools; Test type: Superiority; p = 0.52, Conditional linear regression; Class group as strata. Adjusted for year of birth, sex as well as average temperature, relative humidity and CO2 concentration during the experiment; Relative (percent) changes in the median = 1.37, 95% CI 2-sided [-2.81 to 5.56] — Change comparing the filter group to the non-filter group

2. Primary Outcome: Combined Risk Taking Score
Description: The "Combined risk taking score" measures how willing the person is to take risks and is calculated as 0.4729985 × "Risk preference score" + 0.5270015 × "Willingness to take risks", as defined in Falk et al (2018). The "Combined risk taking score" is a weighted average of two z-scores ("risk preference score" and "willingness to take risks" score), and therefore it can be interpreted as a z-score. The central value of "Combined risk taking score" is 0 and represents the population mean. The higher the values of the "Combined risk taking score", the more willing is the person to take risks. The "Risk preference score" is the final node in the risk tree (see the online appendix of Falk et al (2018)), which is a value between 1 and 32, ranked by the level of risk aversion, which was then transformed to a z-score. The "Willingness to take risks" refers to the answer to the question on one's willingness to take risks, with values from 0 to 10), which was then transformed to a z-score.
Time Frame: Obtained from a test administered approximately 100 minutes after entering the classroom
Measure: Median (Inter-Quartile Range); unit: Z-score
Arm/Group | Purified Air | Normal Air
Number analyzed (Participants) | 1068 | 1054
Z-score | -0.0210 [-0.4730 to 0.4552] | -0.0121 [-0.4580 to 0.4738]
Statistical Analysis 1: Comparison: Purified Air vs Normal Air; The hypothesis was that air filtration could result in higher riskloving behavior, relative to the classroom without air filter (normal air), in the combined risk taking measures among adolescents in high schools; Test type: Superiority; p = 0.72, Regression, Linear; Using multiple imputation by chained equations. Adjusted for a rich set or relevant controls. Standard errors clustered at the high school level; Beta coefficient = 0.013, 95% CI 2-sided [-0.0607 to 0.0865] — Change comparing the filter group to the non-filter group

3. Primary Outcome: Combined Patience Score
Description: The "Combined patience score" measures the patience of the person and is calculated as 0.7115185 × "Time preference score" + 0.2884815 × "Self assessment of patience", as defined in Falk et al (2018). The "Combined patience score" is a weighted average of two z-scores ("time preference score" and "self assessment of patience" score), and therefore it can be interpreted as a z-score. The central value of "Combined patience score" is 0 and represents the population mean. The higher the values of the "Combined patience score" the more patience the person has. The "Time preference score" was obtained from the final node in the time tree (see the online appendix of Falk et al (2018)), which is a value between 1 and 32, ranked by the level of patience, which was then transformed to a z-score. The "Self assessment of patience" score refers to the answer to the question on the self-assessment of patience, with values from 0 to 10, which was then transformed to a z-score.
Time Frame: Obtained from a test administered approximately 100 minutes after entering the classroom
Measure: Median (Inter-Quartile Range); unit: Z-score
Arm/Group | Purified Air | Normal Air
Number analyzed (Participants) | 1068 | 1054
Z-score | -0.1453 [-0.6474 to 0.6330] | -0.0732 [-0.6516 to 0.6575]
Statistical Analysis 1: Comparison: Purified Air vs Normal Air; The hypothesis was that air filtration could result in higher level of patience, relative to the classroom without air filter (normal air), in the combined patience measures among adolescents in high schools; Test type: Superiority; p = 0.50, Regression, Linear; [statistical method as in outcome 2, analysis 1]; Beta coefficient = -0.029, 95% CI 2-sided [-0.1170 to 0.0584] — Change comparing the filter group to the non-filter group

4. Primary Outcome: Positive Reciprocity Score
Description: The "Positive reciprocity score" measures positive reciprocity. A person with high reciprocity agrees with the statement "When someone does me a favor, I am willing to return it". The score is calculated as 0.4847038 × "Willingness to return favor" + 0.5152962 × "Size of gift", as defined in Falk et al (2018). The "Positive reciprocity score" is a weighted average of two z-scores ("willingness to return a favor" score and "size of gift" score), and therefore it can be interpreted as a z-score, with the central value of 0 representing the population mean. Higher values of the score imply more positive reciprocity. "Willingness to return favor" refers to the answer to the question on the willingness to return a favor, ranked from 0 to 10 and then transformed to a z-score. "Size of gift" refers to the answer to the question on the reported size of the gift that would return to a stranger, from a list of 7 possible values (from 0 to 30€, by 5€ steps), then transformed to a z-score.
Time Frame: Obtained from a test administered approximately 100 minutes after entering the classroom
Measure: Median (Inter-Quartile Range); unit: Z-score
Arm/Group | Purified Air | Normal Air
Number analyzed (Participants) | 1068 | 1054
Z-score | -0.0186 [-0.3644 to 0.5352] | -0.0359 [-0.5999 to 0.5372]
Statistical Analysis 1: Comparison: Purified Air vs Normal Air; The hypothesis was that air filtration could result in higher level of positive reciprocity behavior, relative to the classroom without air filter (normal air), in the positive reciprocity measures among adolescents in high schools; Test type: Superiority; p = 0.13, Regression, Linear; [statistical method as in outcome 2, analysis 1]; Beta coefficient = 0.060, 95% CI 2-sided [-0.0184 to 0.1394] — Change comparing the filter group to the non-filter group

5. Primary Outcome: Altruism Score
Description: The "Altruism score" measures the altruism of a person and is calculated as 0.6350048 × "Willingness to give to good causes" + 0.3649952 × "Hypothetical donation", as defined in Falk et al (2018). The "Altruism score" is a weighted average of two z-scores ("willingness to give to good causes" score and "hypothetical donation" score), and therefore it can be interpreted as a z-score, with the central value of 0 representing the population mean. Higher values of the score imply more altruism. "Willingness to give to good causes" refers to the answer to the question on the willingness to give to good causes, ranked from 0 to 10 and then transformed to a z-score. "Hypothetical donation" refers to the answer to the question on the size of the hypothetical donation one would be willing to make, transformed to a z-score.
Time Frame: Obtained from a test administered approximately 100 minutes after entering the classroom
Measure: Median (Inter-Quartile Range); unit: Z-score
Arm/Group | Purified Air | Normal Air
Number analyzed (Participants) | 1068 | 1054
Z-score | 0.1118 [-0.5652 to 0.6197] | 0.0597 [-0.6023 to 0.6754]
Statistical Analysis 1: Comparison: Purified Air vs Normal Air; The hypothesis was that air filtration could result in higher Altruism behavior, relative to the classroom without air filter (normal air), in the Altruism measures among adolescents in high schools; Test type: Superiority; p = 0.58, Regression, Linear; [statistical method as in outcome 2, analysis 1]; Beta coefficient = 0.022, 95% CI 2-sided [-0.0595 to 0.1035] — Change comparing the filter group to the non-filter group

6. Primary Outcome: Trust Score
Description: Answer to the question "I assume that people have only the best intentions", which is ranked from 0 to 10. Higher values imply more trust.
Time Frame: Obtained from a test administered approximately 100 minutes after entering the classroom
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Purified Air | Normal Air
Number analyzed (Participants) | 1068 | 1054
score on a scale | 5 [4 to 7] | 5 [4 to 7]
Statistical Analysis 1: Comparison: Purified Air vs Normal Air; The hypothesis was that air filtration could result in higher trust, relative to the classroom without air filter (normal air), in the subjective trust measure among adolescents in high schools; Test type: Superiority; p = 0.89, Ordered logistic regression; [statistical method as in outcome 2, analysis 1]; Beta coefficient = 0.013, 95% CI 2-sided [-0.1786 to 0.2049] — Change comparing the filter group to the non-filter group

7. Secondary Outcome: Impulsivity (From ANT)
Description: Number of incorrect responses (responses made in the opposite direction to the direction of the target arrow) Lower score indicates a better attention performance. Total range score: 0-38.
Time Frame: Obtained from a test administered approximately 90 minutes after entering the classroom
Measure: Median (Inter-Quartile Range); unit: total score
Arm/Group | Purified Air | Normal Air
Number analyzed (Participants) | 999 | 994
total score | 2 [1 to 4] | 2 [1 to 4]
Statistical Analysis 1: Comparison: Purified Air vs Normal Air; Test type: Superiority; p = 0.50, Conditional linear regression; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.13, 95% CI 2-sided [-0.49 to 0.24] — Change comparing the filter group to the non-filter group

8. Secondary Outcome: Selective Attention (From ANT)
Description: Number of omission errors (failure to respond) Lower score indicates a better attention performance Total range score: 0-21. Higher values represent a worse outcome
Time Frame: Obtained from a test administered approximately 90 minutes after entering the classroom
Measure: Median (Inter-Quartile Range); unit: total score
Arm/Group | Purified Air | Normal Air
Number analyzed (Participants) | 999 | 994
total score | 0 [0 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Purified Air vs Normal Air; Test type: Superiority; p = 0.47, Conditional linear regression; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.20 to 0.10] — Change comparing the filter group to the non-filter group

9. Secondary Outcome: Alerting Score (From ANT)
Description: Alerting represents the ability to maintain a state of high vigilance to incoming stimuli It is calculated by subtracting the median reaction time for double cue from median reaction time for the no cue condition (calculations performed after removing the incongruent trials). A lower score indicates a better attention performance
Time Frame: Obtained from a test administered approximately 90 minutes after entering the classroom
Measure: Median (Inter-Quartile Range); unit: ms
Arm/Group | Purified Air | Normal Air
Number analyzed (Participants) | 999 | 994
ms | 42 [18 to 68.5] | 44.5 [17 to 73]
Statistical Analysis 1: Comparison: Purified Air vs Normal Air; Test type: Superiority; p = 0.20, Conditional linear regression; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.38, 95% CI 2-sided [-8.51 to 1.74]

10. Secondary Outcome: Orienting Score (From ANT)
Description: Orienting is the ability to select information and it is calculated by subtracting the median reaction time for spatial cue from the reaction time for central cue (calculations performed after removing the incongruent trials).A lower score indicates a better attention performance
Time Frame: Obtained from a test administered approximately 90 minutes after entering the classroom
Measure: Median (Inter-Quartile Range); unit: ms
Arm/Group | Purified Air | Normal Air
Number analyzed (Participants) | 999 | 994
ms | 12.5 [-11.5 to 39] | 13.5 [-11.5 to 37.5]
Statistical Analysis 1: Comparison: Purified Air vs Normal Air; Test type: Superiority; p = 0.92, Conditional linear regression; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.25, 95% CI 2-sided [-5.10 to 4.60]

11. Secondary Outcome: Conflict Score (Executive Attention) (From ANT)
Description: Conflict generally refers to the ability to monitor and resolve conflict among responses and in this study it is calculated as the median reaction time for each flanker condition (across cue conditions) and subtracting the congruent from the incongruent reaction times. A lower score indicates a better attention performance
Time Frame: Obtained from a test administered approximately 90 minutes after entering the classroom
Measure: Median (Inter-Quartile Range); unit: ms
Arm/Group | Purified Air | Normal Air
Number analyzed (Participants) | 999 | 994
ms | 75 [57.5 to 93.5] | 75 [58 to 95.5]
Statistical Analysis 1: Comparison: Purified Air vs Normal Air; Test type: Superiority; p = 0.46, Conditional linear regression; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.36, 95% CI 2-sided [-4.94 to 2.22]

12. Secondary Outcome: Self Assessment of How Good They Are in Math
Description: Answer to the question on math skills, ranging from 0 to 10. The higher the score, the better the person feels s/he is doing in math.
Time Frame: Obtained from a test administered approximately 100 minutes after entering the classroom
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Purified Air | Normal Air
Number analyzed (Participants) | 746 | 767
score on a scale | 6 [3 to 8] | 6 [3 to 8]
Statistical Analysis 1: Comparison: Purified Air vs Normal Air; The hypothesis was that air filtration could result in higher assessment of math skills, relative to the classroom without air filter (normal air), in the self assessed math skills measure among adolescents in high schools; Test type: Superiority; p = 0.232, Ordered logistic regression; Adjusted for a rich set or relevant controls. Standard errors clustered at the high school level; Beta coefficient = -0.1446, 95% CI 2-sided [-0.3820 to 0.0928] — Change comparing the filter group to the non-filter group

ADVERSE EVENTS:
Description: Death, serious adverse events and other (non-serious adverse events) were not assessed for the study.
Arm/Group | Purified Air | Normal Air
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-11-20): https://cdn.clinicaltrials.gov/large-docs/39/NCT03762239/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-20): https://cdn.clinicaltrials.gov/large-docs/39/NCT03762239/SAP_001.pdf